CLINICAL TRIAL: NCT00966082
Title: RCT Comparing the Efficacies of Endoscopic Band Ligation (EBL) and Combined Treatment of Beta-blocker and EBL for the Prevention of Esophageal Variceal Rebleeding in Patients With Previous Endoscopic Variceal Treatment
Brief Title: EBL Versus EBL and Propranolol for the Prevention of Variceal Rebleeding in Pts With Previous Variceal Treatment
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Korea University (Other)
Responsible Party: Principal Investigator, Soon Ho Um, Professor, Korea University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EBLPPL-2
Record Dates: First submitted 2009-08-25; First posted 2009-08-26 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Cirrhosis; Variceal Bleeding
Keywords: Cirrhosis; Esophagus Disorders; Varicose Veins
MeSH Terms: conditions — Fibrosis; Esophageal Diseases; Varicose Veins

STUDY DESIGN:
Intervention Model Description: Endoscopic Band Ligation (EBL) Versus Endoscopic Band Ligation and Propranolol
Oversight: Data Monitoring Committee: No

ARMS (2):
- Endoscopic band ligation (Active Comparator): Perform endoscopic band ligation (EBL) until eradication of esophageal varices, and then follow-up endoscopy with 3-6 months interval
  Interventions: Procedure: endoscopic band ligation
- endoscopic band ligation+Propranolol (Active Comparator): Perform endoscopic band ligation (EBL) until eradication of esophageal varices, and then follow-up endoscopy with 3-6 months interval, with propranolol
  Interventions: Procedure: endoscopic band ligation+Propranolol

INTERVENTIONS:
Procedure: endoscopic band ligation — Perform EBL until esophageal varices are eradicated, and then follow-up endoscopy with 3-6 months interval
  Arms: Endoscopic band ligation
Procedure: endoscopic band ligation+Propranolol — Perform EBL same as EBL group. In addition, take propranolol to reduce 25% in HR or HR ≤55/min
  Arms: endoscopic band ligation+Propranolol

SUMMARY:
This study is performed to compare the efficacy and safety of EBL alone and EBL combined with propranolol in patients who were previously performed endoscopic variceal treatment.

DETAILED DESCRIPTION:
Both propranolol and endoscopic band ligation (EBL) are effective for prevention of variceal rebleeding. Recently several studies compared the efficacy of EBL alone and with a combination of propranolol and EBL. However, the results of recent studies showed discrepancy. In addition, most of all recent studies included patients without previous endoscopic treatment for varices. This study is performed to compare the efficacy and safety of EBL alone and EBL combined with propranolol in patients who were previously performed endoscopic variceal treatment.

ELIGIBILITY:
Inclusion Criteria:

* Liver cirrhosis
* Age between 18 and 70 years
* Successful control of esophageal variceal bleeding within 6 weeks before enrollment

Exclusion Criteria:

* Gastric variceal bleeding
* Patients with systolic blood pressure <100 mmHg or basal heart rate <60/min
* Portal vein thrombosis
* Prominent hepatic encephalopathy
* Coexisting untreated malignancy
* Severe cerebrovascular or cardiovascular disease, renal failure
* No previous history of endoscopic, radiologic, or surgical treatment for varices or ascites
* Contraindication to beta-blocker
* Pregnancy
* Refusal to give consent to participate in the trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2008-08; Primary Completion 2019-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Rebleeding from esophageal varices | 2 years
  Rebleeding from esophageal varices

SECONDARY OUTCOMES:
Upper gastrointestinal bleeding; Significant esophageal variceal bleeding; Mortality; Adverse events | 2 years
  Upper gastrointestinal bleeding; Significant esophageal variceal bleeding; Mortality; Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Soon Ho Um, Prof, Principal Investigator — Korea University
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea